CLINICAL TRIAL: NCT01206829
Title: Hearing Impairment, Tinnitus, Mental Health and Vocational Coping. A Randomized, Controlled Study of a Cognitive Therapy Program to Reduce Social Safety Seeking.
Brief Title: Hearing Impairment, Cognitive Therapy and Coping
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); National Centre for Hearing Impairment and Mental Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/2156 (REK); 52-2009 AUS (Other: Kompetansesenter for personvern og sikkerhet, OUS)
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2013-06-14 (Estimated); Status verified 2013-06

CONDITIONS: Hearing Loss; Tinnitus; Stress, Psychological; Mental Fatigue
Keywords: Hearing Impaired Persons; Tinnitus; Life Change Events; Adaptation, Psychological; Rehabilitation, Vocational; Cognitive Therapy; Avoidance Learning; Escape Reaction
MeSH Terms: conditions — Hearing Loss; Tinnitus; Stress, Psychological; Mental Fatigue; Escape Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Audiological rehabilitation (Active Comparator): 16 hours of psychosocial rehabilitation course
  Interventions: Behavioral: 8-session CBTcourse; Behavioral: 8 session cognitive behavioral therapy

INTERVENTIONS:
Behavioral: 8-session CBTcourse — Hearing impaired workers voluntarily sign up for an 8 session cognitive therapy course. The study has a waiting list control group design. Participants will be randomized assigned to either an experiment group that will be offered to start on an immediate course, or a control group that will be offered the same course 12 months later.
Behavioral: 8 session cognitive behavioral therapy — 8 sessions cognitive behavioral therapy in group

SUMMARY:
A randomized controlled study with hearing impaired workers, who have voluntarily signed up for an 8 session cognitive therapy (CBT) course The CBT intervention will be compared to a waiting list control group. Participants who are allocated to the intervention group will be offered to start on the CBT-course immediately, while the control group that will be offered the same course 12 months later. Main outcome measures are assessments of mental distress and vocational coping. We will also assess the distress associated with tinnitus, which is a potential moderator variable.

DETAILED DESCRIPTION:
Although the relationship between hearing loss and mental distress is not linear, it is known that hearing impaired individuals have increased vulnerability for development of symptoms of distress and fatigue. It is assumed that distressed hearing impaired individuals will have a tendency to use maladaptive and passive coping strategies, such as social withdrawal or reluctance to make use of hearing aid devices. On the other side, it is well documented that hearing impaired employers who are open about their handicap and make others aware of their situation, i.e. take an active coping approach, have fewer symptoms of distress and have better vocational functioning. The level of knowledge is limited and mainly based on cross sectional studies, and the way people cope with hearing impairment has been measured indirectly by questionnaires focusing on communication problems. We plan to conduct a randomized controlled study with hearing impaired workers, who have voluntarily signed up for an 8 session cognitive therapy (CBT) course The CBT intervention will be compared to a waiting list control group. Participants who are allocated to the intervention group will be offered to start on the CBT-course immediately, while the control group that will be offered the same course 12 months later. Main outcome measures are assessments of mental distress and vocational coping. We will also assess the distress associated with tinnitus, which is a potential moderator variable.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants need to be within the age range of 18-70 years, contain some formal employment and be able to document a mean, bilateral hearing loss of at least 40 dB.
* Eligible participants need to have a HAD score of 7 or beyond

Exclusion Criteria:

* Individuals without a clear vocational status (for instance on permanent/temporarily sick leave) and a mean bilateral hearing loss beneath 40 dB.
* Individuals with a HAD score beneath 8 are excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Work Ability Index | At recruitment, at time of course completement and at 6 months post-treatment
  Work Ability Index is a self report instrument that measures changes and variations in level of vocational functioning.
Current employment status | At recruitment, at time of course completement and at 6 months post-treatment.
  Participants are asked to desribe their current vocational situation in some more detail. In addition, one item from the General Health Questionnaire, GQH-20 (World Health Organization, 2007) is included here: "To what degree is your ability to perform your ordinary work reduced today?"
Hospital Anxiety and Depression Scale; HADS | At recruitment, at time of course completement and at 6 months post-treatment.
  HADS consists of 14 items covering symptoms of anxiety and depression. HADS is a standarized and validated self report measure of general, mental health.
Fear of Negative Evaluation (FNE) | At recruitment, at time of course completement and at 6 months post-treatment.
  FNE is a self report questionnaire covering symptoms of social phobia. FNE is often used to measure treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Egil W Martinsen, Prof. dr. med., Study Chair — Oslo University Hospital; Katharine C Williams, cand. psychol., Principal Investigator — The Norwegian Centre for Hearing Impairment and Mental Health
Locations (1):
- The Norwegian Centre for Hearing Impairment and Mental Health Oslo University Hospital, Oslo, Norway, Norway